CLINICAL TRIAL: NCT01018589
Title: Effect the Cicatrix Cream in in Treatment of Post Surgical Scars and and Epidermic Burn.
Brief Title: Cicatrix Cream in Post Surgical Scars and Epidermic Burn
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Catalysis SL (Industry)
Responsible Party: Edelisa Moredo Romo, Juan Manuel Marquez Pediatric Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAT-0904-CU
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2010-12-08 (Estimated); Status verified 2010-12

CONDITIONS: Post Surgical Scars; Epidermic Burn
Keywords: Post surgical scars; Epidermic burn; Cicatrix cream

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- A (Experimental): Cicatrix cream
  Interventions: Other: Cicatrix cream

INTERVENTIONS:
Other: Cicatrix cream — We will be carried out the topical application of the product (Cicatrix cream) in the epidermic burns or post surgical scars by administration fo the patients twice a day during two months to a dose of 0,1 ml of cream for each cm of surface, being controlled by the specialist in biweekly consultations.
  To the patient will be explained the technique of the application.

SUMMARY:
The purpose of the study is to assess the effect of CICATRIX (Asian Gotu Kola or Pennywort) usage in the treatment of epidermic burns or post surgical scars. The duration of this phase 2 clinical trial will be two months.

ELIGIBILITY:
Inclusion Criteria:

* Patient with lesions characteristic of the investigated illness.
* Signed informed consent

Exclusion Criteria:

* Patient that refer manifestations of high sensibility to the medication or to some of the components of the product
* Patient that don't want to participate in the study
* Patient not very cooperative
* Family responsible not very cooperative

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Reduction of the areas of lesions at 2 months (end of the treatment) | 2 months

SECONDARY OUTCOMES:
Coloration of the lesions at 2 months (end of the treatment) | 2 months
Adverse effects | 2 months

CONTACTS AND LOCATIONS:
Overall Officials: Edelisa Moredo Romo, MD, Principal Investigator — Juan Manuel Marquez Pediatric Hospital
Locations (1):
- Juan Manuel Marquez Pediatric Hospital, Havana, La Habana, Cuba